CLINICAL TRIAL: NCT05846100
Title: Conventional Palpation Versus Ultrasound Assisted Spinal Anesthesia in Obstetrics: A Randomized Controlled Trial
Brief Title: Conventional Palpation Versus Ultrasound Assisted Spinal Anesthesia in Obstetrics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mongi Slim Hospital (Other)
Responsible Party: Principal Investigator, Mhamed Sami Mebazaa, Conventional palpation versus ultrasound assisted spinal anesthesia in obstetrics: A randomized controlled trial, Mongi Slim Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Ultrasound spinal anesthesia
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Obese; Cesarean Section; Anesthesia Spinal
Keywords: spinal anesthesia; ultrasound; c section
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: All eligible participants scheduled for cesarean delivery were prospectively randomized to 2 groups using computer-generated random numbers:
  A standard manual palpation group (standard group, n=45) and a pre-puncture ultrasound-guided neuraxial anesthesia group (ultrasound group, n=45).
Who Masked: Participant
Masking Description: Fictional ultrasound identification Screen device shut down Intervertebral space identified using the standard palpation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard group (Placebo Comparator): Fictional ultrasound identification Screen device shut down Intervertebral space identified using the standard palpation
  Interventions: Procedure: fictional preprocedure spinal ultrasound
- ultrasound group (Active Comparator): pre-puncture ultrasound-guided neuraxial anesthesia group
  Interventions: Procedure: Preprocedural spinal ultrasound

INTERVENTIONS:
Procedure: Preprocedural spinal ultrasound — a preprocedural spinal ultrasound was performed in a non sterile manner with a sitting position.Both paramedian and transverse planes The intersection of the longitudinal and transverse lines is the point of needle insertion The distance from the skin to the dura mater is noted
  Arms: ultrasound group
Procedure: fictional preprocedure spinal ultrasound — fictional preprocedure spinal ultrasound Fictional ultrasound identification Screen device shut down
  Arms: standard group

SUMMARY:
Spinal anesthesia in obese parturients is commonly difficult yet there are no guidelines to direct best practice. The failure leads to suboptimal patient outcomes.

Ultrasonography is now considered standard care for central venous access and regional anesthesia and it can be used to visualize the anatomy of the spine for this procedure.

Goal of the study

Evaluate the benefits of preprocedural ultrasound scanning to facilitate neuraxial anesthesia and improve the first-attempt success rate in obese parturients.

DETAILED DESCRIPTION:
This was a prospective, randomized controlled trial conducted between Nov 2022 and December 2022 in the gynecological operating room of Mongi Slim hospital.

Ethical approval was provided by our Institutional Hospital Ethics Committee.

Written informed consent was obtained from all the participants.

Study population

1. Inclusion criteria

   * Age >18 years old
   * Normal singleton pregnancy
   * Gestational age ≥ 37 weeks
   * BMI ≥ 30 Kg/ m2 (weight measured on the day before delivery)
   * Planned cesarean section
   * ASA 2-3
2. Non-inclusion criteria

   * Patient refusal to participate or unable to provide consent
   * Emergency cesarean section
   * patient pregnant with twins
   * Contraindications to spinal anesthesia:
   * Localized sepsis: infection at the puncture site
   * allergy to any of the drugs planned fo administration
   * raised intracranial pressure
   * spine surgery
   * aortic stenosis
   * Coagulopathy
   * hypovolemia
3. Exclusion criteria

   * Spinal anesthesia failure
   * Poorly Tolerated spinal anesthesia

Methods

All eligible participants scheduled for cesarean delivery were prospectively randomized to 2 groups using computer-generated random numbers:

A standard manual palpation group (standard group, n=45) and a pre-puncture ultrasound-guided neuraxial anesthesia group (ultrasound group, n=45).

The sample size calculation was based on a previous study [1], the first-attempt success rate was 52% in the conventional approach and 87% in the ultrasound group.

With an α error of 5% and a ß error of 20% (80% power), a sample size of 43 patients per group was required. We increased the number to 45 per group to allow dropouts.

The weight, height and BMI of the parturients were measured one day before the delivery.

The degree of obesity was determined according to the classification of body mass index of the world health organization.

In the operating room, patients were monitored with pulse oximetry, non invasive blood pressure and 3-lead electrocardiogram. Intravenous access was established. Randomization was revealed at this time.

Eligible operators for the study were anesthesia fellows and residents in their third and fourth year of training anesthesia. Fellows and residents received didactic teaching in the form of reading material and educational video on spinal sonography before patient recruitment and were instructed on how to perform a standardized spinal ultrasound assessment for neuraxial procedures. The training proceeded with a demonstration on a live model with typical sonoanatomy at all lumbar spaces and were required to perform the following tasks:

1. identification of the sacrum and five lumbar intervertebral spaces in the paramedian sagittal oblique plane.
2. determination of the midline and the interspace at different lumbar interspaces, the optimal needle insertion point and the distance from the skin to the inner aspect of the ligamentum flavum and dura mater unit in the transverse median plane.

A portable ultrasound system (sonosite) equipped with a curved array probe was utilized.

In the standard group, with the parturient in a sitting position, the anaesthesiologist identified the L4-L5 space using the standard palpation method : the imaginary line connecting both upper iliac crests crossing the spine identified the L4-L5 interspace. The duration required to identify the point of puncture is noted.

In the ultrasound group, a preprocedural spinal ultrasound was performed in a non sterile manner with a sitting position. Ultrasound visualization in both paramedian and

transverse planes was performed. The convex transducer was first placed on the sacral region on a longitudinal paramedian presentation, 2-3cm from the midline, angled to the spinal canal which leads to the identification of the sacrum as a continuous hyperechoic line. Then the transducer was moved in a cephalad direction to identify the intervertebral spaces as acoustic windows and spinous processes as acoustic shadows. We draw a transverse line with a disposable skin marker at either the L3-4 or L4-5 interspace. Then we rotate the probe 90 degrees and place transversely to determine the midline, which was marked by a longitudinal line. The intersection of the longitudinal and transverse lines is the point of needle insertion. We tilt the probe slightly up and down to ensure a sufﬁcient echogenic window at the selected intervertebral level. The distance from the skin to the dura mater is noted.

The time required to identify the insertion site is noted.

In both groups, we record the procedure time which is time from the handle of the spinal needle to observe free flow of cerebrospinal fluid.

After a full aseptic painting, spinal anesthesia was administered using a 25-gauge, 90-mm pencil-point needle inserted through a 20-gauge introducer needle with hyperbaric bupivacaine, 2,5 μg sufentanil and preservative-free morphine 100μg.

The dose of bupivacaine will be selected based on the height of the parturient as shown in the table below (table1).

The patient was positioned supine with left uterine displacement then surgery was allowed to proceed once bilateral sensory block to cold spray to T4 was achieved.

Outcome measures

primary outcome:

-First pass success rate without needle redirection or reinsertion.

Secondary outcomes:

1. Number of puncture attempts : new skin puncture at the same or different interspace
2. Number of intervertebral interspaces attempted
3. Requirement of needle redirection : any withdrawal and re-advancement of the spinal needle and/or introducer within an intervertebral space
4. Procedure Time ( total time required for the identification + time from first placement of the introducer until free flow of cerebrospinal fluid.
5. Patient satisfaction score.
6. Possible complications:

   * Traumatic procedure
   * Postdural puncture headache
   * Development of back pain post spinal anesthesia
   * paresthesia

Ethical Considerations:

All patients were included after obtaining their informed consent (Appendix).

Participation was voluntary and anonymous.

We explained to the participants:

* The usefulness of this study
* Absence of significant adverse effects at this dose (low dose).
* The possibility of accepting or refusing participation.
* The possibility of leaving the study at any time

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* Normal singleton pregnancy
* Gestational age ≥ 37 weeks
* BMI ≥ 30 Kg/ m2 (weight measured on the day before delivery)
* Planned cesarean section
* ASA 2-3

Exclusion Criteria:

* Spinal anesthesia failure
* Poorly Tolerated spinal anesthesia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — OBESE PARTURIENTS
Enrollment: 90 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
First pass success rate | before spinal anesthesia
  First pass success rate without needle redirection or reinsertion

SECONDARY OUTCOMES:
Number of puncture attempts | before spinal anesthesia
  new skin puncture at the same or different interspace
Number of intervertebral interspaces attempted | before spinal anesthesia
Requirement of needle redirection | before spinal anesthesia
  any withdrawal and re-advancement of the spinal needle and/or introducer within an intervertebral space
Procedure Time | before spinal anesthesia
  total time required for the identification + time from first placement of the introducer until free flow of cerebrospinal fluid
Patient satisfaction score | before spinal anesthesia
Possible complications | before spinal anesthesia
  Traumatic procedure
  * Postdural puncture headache
  * Development of back pain post spinal anesthesia
  * paresthesia

CONTACTS AND LOCATIONS:
Overall Officials: Amani BEN HAJ YOUSSEF, Principal Investigator — Mongi Slim local research ethical committee
Locations (1):
- Mongi Slim hospital, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No